CLINICAL TRIAL: NCT02677415
Title: Impact of General vs Local Anesthesia on Neurological Function in Patients With Acute Ischemic Stroke Undergoing Endovascular Treatment
Brief Title: Impact of Anesthesia Type on Outcome in Patients With Acute Ischemic Stroke (AIS) Undergoing Endovascular Treatment
Acronym: CANVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, M.D., Ph.D., Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: QML20150508
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Acute Stroke
Keywords: Ischemic Stroke; Anesthesia; Endovascular Procedures
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Anesthetics, Intravenous; Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anesthesia (Other): local anesthesia and spontaneous breathing will be maintained.
  Interventions: Other: local anesthesia; Other: Spontaneous breathing
- General anesthesia (Other): Intravenous anesthetics and controlled ventilation will be used .
  Interventions: Other: Intravenous anesthetics; Other: Controlled ventilation

INTERVENTIONS:
Other: Intravenous anesthetics
  Arms: General anesthesia
Other: local anesthesia
  Arms: Local anesthesia
Other: Controlled ventilation
  Arms: General anesthesia
Other: Spontaneous breathing
  Arms: Local anesthesia

SUMMARY:
Recent observational studies have found an association between general anaesthesia and increased post-operative mortality in acute ischemic stroke patients undergoing endovascular treatment. It is unknown whether there is a causal relationship in this observation. The investigators are performing a large randomised trial of general versus local anaesthesia to definitively answer the question of whether anaesthetic type alters perioperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AIS scheduled to receive emergency endovascular treatment, older than 18; the onset time is within 12 hours.

Exclusion Criteria:

* Radiological ambiguity concerning infarction and vessel occlusion.
* Additional intracerebral hemorrhage.
* Posterior circulation infraction.
* Coma on admission (Glasgow coma score less than 8).
* NIHSS less than 10 or more than 35.
* Severe agitation or seizures on admission.
* Obvious loss of airway protective reflexes and/or vomiting on admission.
* Being intubated before treatment on admission.
* Known allergy to anesthetic or analgesic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
modified Rankin score | post-procedural 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D., Principal Investigator — Department of Anesthesiology, Beijing Tiantan Hospital
Locations (1):
- Beijing TianTan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Peng Y, Li Y, Jian M, Liu X, Sun J, Jia B, Dong J, Zeng M, Lin N, Zhang L, Gelb AW, Chan MT, Han R. Choice of ANesthesia for EndoVAScular Treatment of Acute Ischemic Stroke: Protocol for a randomized controlled (CANVAS) trial. Int J Stroke. 2017 Dec;12(9):991-997. doi: 10.1177/1747493017706243. Epub 2017 Apr 24. PMID 28436307